CLINICAL TRIAL: NCT03048032
Title: Diagnostic and Prognostic Value of Cardiac Biomarkers and Echocardiography for Patients Hospitalized Due to Acute Dyspnea: Prospective Observational Multicenter Cohort Study
Brief Title: Lithuanian Echocardiography Study of Dyspnea in Acute Settings
Acronym: LEDA
Status: Completed | Type: Observational
Sponsor: Vilnius University (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Jelena Čelutkienė, Senior Researcher and Professor in Clinic of Cardiac and Vascular Diseases, Centre of Cardiology and Angiology, Vilnius University; Senior cardiologist in Unit of Stress testing, Vilnius University hospital Santariškių Klinikos, Vilnius University
Other Study IDs: MIP-049/2015; MIP-049/2015 (Other Grant/Funding Number: Research Council of Lithuania); L-15-01/1 (Other: Lithuanian Bioethics Commitee)
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Acute Heart Failure
Keywords: acute heart failure; right ventricular failure; cardiac biomarkers; echocardiography; diagnosis; prognosis
MeSH Terms: conditions — Heart Failure; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute heart failure patients: Adult patients (18 years and older) who are admitted to the emergency department (Vilnius University Hospital Santariškių Klinikos and Hospital of Lithuanian University of Health Sciences Kauno Klinikos) due to acute dyspnea and have an adjudicated diagnosis of acute heart failure. Blood sampling and echocardiography examination will be performed.
  Interventions: Procedure: Blood sampling; Procedure: Echocardiography exam
- Control group: Patients who are admitted to the emergency departments of participating centers due to acute dyspnea with an adjudicated diagnosis other than heart failure (pulmonary causes of dyspnea such as pulmonary embolism, acute infections, cancer and other reasons). Blood sampling and echocardiography examination will be performed.
  Interventions: Procedure: Blood sampling; Procedure: Echocardiography exam

INTERVENTIONS:
Procedure: Blood sampling — Besides routine clinical, laboratory and instrumental evaluation, blood samples will be taken within 4 hours of presentation to the hospital. Plasma samples, stored and frozen at -80°C, will be analyzed at the INSERM UMR942 institute in Paris. Up to 15 novel will be measured during the study: copeptine, proenkephalin, high sensitivity troponin T, troponin I, brain natriuretic peptide (BNP), N-terminal pro-BNP, adrenomedullin, soluble ST2, galectine 3, C-reactive protein, interleukine 6, procalcitonin, cystatin C, neutrophil gelatinase associated lipocalin.
Procedure: Echocardiography exam — A standard echocardiography as well as examination focused on right ventricle (RV) will be performed in a period of 48 hours of admission. Novel qualitative and quantitative parameters of right ventricle function and structure will be measured. These include RV diameter at base and midlevel, a measure of RV fractional area change (FAC), tissue doppler imaging derived tricuspid lateral annular systolic velocity wave (S'), tricuspid annular plane systolic excursion (TAPSE), velocity and gradient of tricuspid regurgitation, estimated systolic RV and RA pressure, RV wall strain and strain rate.

SUMMARY:
LEDA (Lithuanian Echocardiography study of Dyspnea in Acute settings) is a prospective observational cohort multicenter clinical study. Project is carried out by Vilnius University together with a partner Lithuanian University of Health Sciences, in conjunction with a research protocol of international GREAT consortium (Global Research on Acute Conditions Team). The aim of this project is to find the specific novel biomarkers of acute heart failure (AHF), to evaluate their diagnostic and prognostic role in association with echocardiographic parameters of AHF. Primary endpoint is 1-year all-cause mortality and rehospitalization. Secondary endpoints are 1) in-hospital all-cause mortality 2) post-discharge 1 and 3 month all-cause mortality and rehospitalization 3) post-discharge 1 and 3 month cardiovascular mortality and rehospitalization 4) one-year cardiovascular mortality and rehospitalization.

During the project a sizeable national database (2000 Lithuanian patients) will be integrated into database of GREAT network. Novel cardiac biomarkers together with ultrasound parameters of right ventricular (RV) function are in the focus of the study. During the acute phase of heart failure, up to 15 novel cardiac, vascular, renal impairment and inflammation biomarkers in plasma samples will be investigated in Lithuania and France (INSERM laboratory). Plasma samples will be taken during 4 hours after admission and frozen at -80ºC to allow batch analysis. The extensive evaluation of innovative ultrasound parameters of right ventricular structure and function will be performed in the early hospitalization period, along with standard echocardiography examination. The first database of AHF patients in Lithuania will provide demographic data and trends of morbidity and mortality, as well as analysis of diagnostic and prognostic value of novel biomarkers and echocardiography parameters in the Baltic region. Quantitative parameters of RV systolic function and deformation will be measured. It is expected that optimal use of novel biomarkers and reproducible echocardiography parameters in the setting of emergency and critical care would reduce unnecessary hospitalizations, cost and hospital length of stay without decrease in the quality of diagnostics and treatment. An estimation of correlation of echocardiographic parameters and biomarkers could help create an accurate algorithm for risk stratification and diagnosis of AHF in an emergency setting.

DETAILED DESCRIPTION:
Heart failure (HF) is believed to be the modern-day epidemic due to increasing incidence, impaired long-term prognosis and huge economic burden. With the ageing population the impact of HF on health care resources is on the rise. The course of the disease is characterized by episodes of acute decompensation that mark a significant turning point in the progress of the disease, with in-hospital mortality rates as high as 10%. Acute heart failure (AHF) is a gradual or rapid change in HF signs and symptoms, requiring urgent medical therapies. Acute heart failure is estimated to be the most costly and the most frequent cause of admission to emergency wards. Emergency department (ED) is the primary setting where initial AHF management takes place. However, strong evidence for diagnostics and management of this grave condition is still lacking. Even less is known about the prevalence, diagnosis and management of acute right ventricular failure (RVF).

A patient presenting to the ED with acute dyspnea has to undergo numerous procedures in order to differentiate the diagnosis between AHF, chronic obstructive pulmonary disease, pneumonia, pulmonary embolism and other etiologies. Moreover, the majority of HF patients suffer from comorbidities that make the diagnostic process even more challenging. Due to numerous exams and tests, the initial management of these patients may be delayed, resulting in an extended hospital length of stay, increased rate of complications and death. The clinical, hemodynamic and neurohormonal features of heart failure are diﬀerent in specific patient populations and depend on age, sex, race, left ventricular ejection fraction and co-existent right ventricular (RV) dysfunction as well as many other factors.

Cardiac biomarkers are easily reproducible and objective laboratory tests that could help to improve early AHF diagnosis and risk stratification. However, reported data suggest varying prognostic and diagnostic values of natriuretic peptides, such as N-type natriuretic peptide (BNP), N-terminal pro B-type natriuretic peptide (NT-proBNP), MR pro-atrial natriuretic peptide (MR-proANP), as well as regional differences of these markers. Specific biomarkers of RVF have not yet been described, thus a search of novel serologic markers that could rapidly and reliably help diagnose acute RVF is a very important scientific task in cardiology. Furthermore, the knowledge on the incidence of RVF syndrome as well as the diagnostic and prognostic values of ultrasound RV structural and functional parameters is scarce. During this study the RV-focused ultrasound examination will be performed in the early hospitalization period, and blood samples will be taken and frozen at the same time. Up to 15 novel cardiac, vascular, renal impairment and inflammation biomarkers in plasma samples during acute phase of RVF will be investigated during the study in France, INSERM laboratory. The study will be unique as it will aggregate large scale observational and biomarkers database of AHF patients in Lithuania together with innovative ultrasound parameters of RV failure (quantitative parameters of RV systolic function and deformation).

The aim of this project is to find the specific novel biomarkers of acute heart failure (AHF), to evaluate their diagnostic and prognostic role in association with echocardiographic parameters of AHF.

The primary endpoint is 1-year all-cause mortality and rehospitalization.

Secondary endpoints are:

1. in-hospital all-cause mortality
2. post-discharge 1 and 3 months all-cause mortality and rehospitalization
3. post-discharge 1 and 3 months cardiovascular mortality and rehospitalization
4. one-year cardiovascular mortality and rehospitalization.

Objectives of this project are:

1. To create a database of patients hospitalized due to acute heart failure in Lithuania, integrated to GREAT (Global Research on Acute Conditions Team) network database;
2. To compare the diagnostic and prognostic value of novel cardiac, vascular, renal insuﬃciency and inflammation biomarkers in the Lithuanian patient cohort to other countries in the GREAT network;
3. To determine the demographic, clinical and treatment characteristics as well as short and long term outcome of patients hospitalized due to AHF in Lithuania and other GREAT network countries;
4. To evaluate the epidemiology of RVF together with clinical features and outcome of patients in a cohort of Lithuanian acute heart failure (HF) patients;
5. To estimate a correlation between ultrasound parameters of RV structure and function and novel cardiac, vascular, renal and inflammation biomarkers in acute period of HF;
6. To identify novel ultrasound parameters of RV structure and function parameters and biomarkers predicting a risk of 1 year mortality after hospitalization;
7. To create an algorithm of RV failure diagnostics and risk stratification based on the diagnostic and prognostic value of detected echocardiographic parameters and biomarkers.

Observational studies and recent meta-analyses indicate that in acute conditions RVF may be as frequent as let ventricular failure (LVF) and is associated with markedly poor prognosis. Largely empiric knowledge in emergency medicine suggests that right and left ventricular failure requires diﬀerent therapeutic approaches, including disparate principles of intravenous treatment, due to distinct hemodynamic impairment. The outcome of RVF is largely dependent on the underlying cause, resulting in either an acute or chronic presentation.

Novel biomarkers can help identify the underlying conditions in AHF. These include myocardial injury markers such as copeptine, proenkephalin, high sensitivity troponin T, troponin I, brain natriuretic peptide (BNP), N-terminal-proBNP; renal and hepatic involvement markers such as adrenomedullin, neutrophil gelatinase-associated lipocalin (NGAL), L-type fatty acid binding protein (L-FABP), galectin-3, soluble ST2, cystatin C; inflammatory markers such as C-reactive protein, interleukine 6, procalcitonin. These markers could help evaluate end-organ involvement, as well as the extent of myocardial remodeling, and in return provide state-of-the-art tailored patient care. Specific biomarkers of RV involvement or dysfunction have not yet been described, therefore identification of such biomarkers would allow to accelerate the diagnosis of RVF and initiate specific treatment.

Echocardiography is a potent and accessible technique for the diagnosis of AHF in an acute setting. Echocardiography also provides information about the mechanisms of AHF as well as alternative causes of dyspnea. Echocardiographic parameters of RV structure and function are of particular interest since not much data is available on acute RVF. Quantitative parameters of RV systolic and diastolic function, RV wall deformation or notional hemodynamic parameters could potentially be useful for diagnosis and selection of urgent treatment tactics. In the current literature there are no publications about the diagnostic and prognostic value of RV parameters, especially about novel echocardiographic parameters (strain rate, speckle tracking), in the early phase of exacerbated heart failure.

Global Research on Acute Conditions Teal (GREAT) Association is an international network among experts operating in the management of acute clinical conditions in the field of emergency medicine and doing research through the concept of translational medicine. This network integrates research inputs from basic sciences and interventional epidemiology to optimize both patient care and preventive measures. Moreover, one of the main objectives of the GREAT association is to standardize the clinical and organizational system approach in acute conditions disease management all over the world, with the concept of globalization medicine. Up to this day there has not been any large multicenter observational and biomarkers studies in Lithuania in the field of AHF. Our study creates a unique opportunity to join the worldwide GREAT network and its patient database, that could potentially contain up to 50 000 patients.

ELIGIBILITY:
Inclusion Criteria:

* presentation to hospital with acute dyspnea.

Exclusion Criteria:

* refusal to give informed consent; acute coronary syndromes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years and older) who present to the hospital (Vilnius University hospital Santariškių Klinikos and Hospital of Lithuanian University of Health Sciences Kauno Klinikos) due to acute dyspnea. Besides acute heart failure, patients with pulmonary causes of dyspnea as well as pulmonary embolism, acute infections, cancer and other reasons are enrolled. Patients admitted to the ward as well as and discharged home from the emergency department are enrolled.
Sampling Method: Probability Sample
Enrollment: 1566 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
1-year all-cause mortality and rehospitalization | 1 year
  The sum of all-cause deaths and all-cause rehospitalizations in AHF and non-AHF groups

SECONDARY OUTCOMES:
In-hospital all-cause mortality | 28 days
  All-cause deaths before discharge in AHF and non-AHF groups
Post-discharge all-cause mortality and rehospitalization | 1 and 3 months
  The sum of all-cause deaths and all-cause rehospitalizations in AHF and non-AHF groups in 1 and 3 months minus Outcome 2
Post-discharge cardiovascular mortality and rehospitalization | 1 and 3 months
  The sum of cardiovascular deaths and cardiovascular rehospitalizations in AHF and non-AHF groups in 1 and 3 months minus Outcome 2
1-year cardiovascular mortality and rehospitalization | 1 year
  The sum of cardiovascular deaths and cardiovascular rehospitalizations in AHF and non-AHF groups

OTHER OUTCOMES:
Prognostic role of circulating biomarkers | 1 year
  Hazard ratio and odds ratio of NT-proBNP, GDF-15 and troponin for primary and secondary outcomes
Prognostic role of echocardiographic parameters | 1 year
  Hazard ratio and odds ratio of TAPSE, LVEF, RV strain for primary and secondary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jelena Celutkiene, Professor, Study Chair — Vilnius University; Ausra Kavoliuniene, Professor, Principal Investigator — Lithuanian University of Health Sciences; Alexandre Mebazaa, Professor, Principal Investigator — INSERM, BIOmarkers in CArdioNeuroVAScular diseases
Locations (3):
- Inserm U942, Paris, Île-de-France Region, France
- Lithuania (2):
  - Lithuanian University of Health Sciences, Kaunas
  - Vilnius University, Vilnius

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to other researchers via GREAT (Global REsearch on Acute Conditions Team) database
Supporting Information: Study Protocol
Time Frame: 2019-2024
Access Criteria: referral to prof. A. Mebazaa

REFERENCES:
- [Background] Kaur M, Sprague S, Ignacy T, Thoma A, Bhandari M, Farrokhyar F. How to optimize participant retention and complete follow-up in surgical research. Can J Surg. 2014 Dec;57(6):420-7. doi: 10.1503/cjs.006314. No abstract available. PMID 25421086
- [Background] Lasagna L. Problems in publication of clinical trial methodology. Clin Pharmacol Ther. 1979 May;25(5 Pt 2):751-3. doi: 10.1002/cpt1979255part2751. PMID 373967
- [Background] Gullen WH, Bearman JE, Calvert JC, Loewenson RB. Medical statistics: unscrambling the clinical research egg. Patient Care. 1978 May 30;12(10):120-2, 127, 130-2 passim. No abstract available. PMID 10236742
- [Background] Julious SA, Owen RJ. Sample size calculations for clinical studies allowing for uncertainty about the variance. Pharm Stat. 2006 Jan-Mar;5(1):29-37. doi: 10.1002/pst.197. PMID 17080926
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Zannad F, Mebazaa A, Juilliere Y, Cohen-Solal A, Guize L, Alla F, Rouge P, Blin P, Barlet MH, Paolozzi L, Vincent C, Desnos M, Samii K; EFICA Investigators. Clinical profile, contemporary management and one-year mortality in patients with severe acute heart failure syndromes: The EFICA study. Eur J Heart Fail. 2006 Nov;8(7):697-705. doi: 10.1016/j.ejheart.2006.01.001. Epub 2006 Mar 3. PMID 16516552
- [Background] Maisel AS, Peacock WF, McMullin N, Jessie R, Fonarow GC, Wynne J, Mills RM. Timing of immunoreactive B-type natriuretic peptide levels and treatment delay in acute decompensated heart failure: an ADHERE (Acute Decompensated Heart Failure National Registry) analysis. J Am Coll Cardiol. 2008 Aug 12;52(7):534-40. doi: 10.1016/j.jacc.2008.05.010. PMID 18687247
- [Background] Emerman CL. Treatment of the acute decompensation of heart failure: efficacy and pharmacoeconomics of early initiation of therapy in the emergency department. Rev Cardiovasc Med. 2003;4 Suppl 7:S13-20. PMID 14668696
- [Background] Peacock WF, Emerman C, Costanzo MR, Diercks DB, Lopatin M, Fonarow GC. Early vasoactive drugs improve heart failure outcomes. Congest Heart Fail. 2009 Nov-Dec;15(6):256-64. doi: 10.1111/j.1751-7133.2009.00112.x. PMID 19925503
- [Background] Masip J, Roque M, Sanchez B, Fernandez R, Subirana M, Exposito JA. Noninvasive ventilation in acute cardiogenic pulmonary edema: systematic review and meta-analysis. JAMA. 2005 Dec 28;294(24):3124-30. doi: 10.1001/jama.294.24.3124. PMID 16380593
- [Background] Maisel AS, McCord J, Nowak RM, Hollander JE, Wu AH, Duc P, Omland T, Storrow AB, Krishnaswamy P, Abraham WT, Clopton P, Steg G, Aumont MC, Westheim A, Knudsen CW, Perez A, Kamin R, Kazanegra R, Herrmann HC, McCullough PA; Breathing Not Properly Multinational Study Investigators. Bedside B-Type natriuretic peptide in the emergency diagnosis of heart failure with reduced or preserved ejection fraction. Results from the Breathing Not Properly Multinational Study. J Am Coll Cardiol. 2003 Jun 4;41(11):2010-7. doi: 10.1016/s0735-1097(03)00405-4. PMID 12798574
- [Background] Januzzi JL Jr, Camargo CA, Anwaruddin S, Baggish AL, Chen AA, Krauser DG, Tung R, Cameron R, Nagurney JT, Chae CU, Lloyd-Jones DM, Brown DF, Foran-Melanson S, Sluss PM, Lee-Lewandrowski E, Lewandrowski KB. The N-terminal Pro-BNP investigation of dyspnea in the emergency department (PRIDE) study. Am J Cardiol. 2005 Apr 15;95(8):948-54. doi: 10.1016/j.amjcard.2004.12.032. PMID 15820160
- [Background] Peacock WF 4th, De Marco T, Fonarow GC, Diercks D, Wynne J, Apple FS, Wu AH; ADHERE Investigators. Cardiac troponin and outcome in acute heart failure. N Engl J Med. 2008 May 15;358(20):2117-26. doi: 10.1056/NEJMoa0706824. PMID 18480204
- [Background] Logeart D, Isnard R, Resche-Rigon M, Seronde MF, de Groote P, Jondeau G, Galinier M, Mulak G, Donal E, Delahaye F, Juilliere Y, Damy T, Jourdain P, Bauer F, Eicher JC, Neuder Y, Trochu JN; Heart Failure of the French Society of Cardiology. Current aspects of the spectrum of acute heart failure syndromes in a real-life setting: the OFICA study. Eur J Heart Fail. 2013 Apr;15(4):465-76. doi: 10.1093/eurjhf/hfs189. Epub 2012 Nov 27. PMID 23186936
- [Background] Chioncel O, Ambrosy AP, Bubenek S, Filipescu D, Vinereanu D, Petris A, Christodorescu R, Macarie C, Gheorghiade M, Collins SP; Romanian Acute Heart Failure Syndromes study investigators. Epidemiology, pathophysiology, and in-hospital management of pulmonary edema: data from the Romanian Acute Heart Failure Syndromes registry. J Cardiovasc Med (Hagerstown). 2016 Feb;17(2):92-104. doi: 10.2459/JCM.0000000000000192. PMID 25252041
- [Background] Belohlavek J, Dytrych V, Linhart A. Pulmonary embolism, part I: Epidemiology, risk factors and risk stratification, pathophysiology, clinical presentation, diagnosis and nonthrombotic pulmonary embolism. Exp Clin Cardiol. 2013 Spring;18(2):129-38. PMID 23940438
- [Background] Kinch JW, Ryan TJ. Right ventricular infarction. N Engl J Med. 1994 Apr 28;330(17):1211-7. doi: 10.1056/NEJM199404283301707. PMID 8139631
- [Background] Naeije R, Brimioulle S, Dewachter L. Biomechanics of the right ventricle in health and disease (2013 Grover Conference series). Pulm Circ. 2014 Sep;4(3):395-406. doi: 10.1086/677354. PMID 25621153
- [Background] Berlin DA, Bakker J. Understanding venous return. Intensive Care Med. 2014 Oct;40(10):1564-6. doi: 10.1007/s00134-014-3379-4. Epub 2014 Jun 26. No abstract available. PMID 24966066
- [Background] Haddad F, Couture P, Tousignant C, Denault AY. The right ventricle in cardiac surgery, a perioperative perspective: I. Anatomy, physiology, and assessment. Anesth Analg. 2009 Feb;108(2):407-21. doi: 10.1213/ane.0b013e31818f8623. PMID 19151264
- [Background] Markel TA, Wairiuko GM, Lahm T, Crisostomo PR, Wang M, Herring CM, Meldrum DR. The right heart and its distinct mechanisms of development, function, and failure. J Surg Res. 2008 May 15;146(2):304-13. doi: 10.1016/j.jss.2007.04.003. Epub 2007 Nov 26. PMID 18036544
- [Background] Mullens W, Abrahams Z, Francis GS, Sokos G, Taylor DO, Starling RC, Young JB, Tang WHW. Importance of venous congestion for worsening of renal function in advanced decompensated heart failure. J Am Coll Cardiol. 2009 Feb 17;53(7):589-596. doi: 10.1016/j.jacc.2008.05.068. PMID 19215833
- [Background] Lankeit M, Jimenez D, Kostrubiec M, Dellas C, Hasenfuss G, Pruszczyk P, Konstantinides S. Predictive value of the high-sensitivity troponin T assay and the simplified Pulmonary Embolism Severity Index in hemodynamically stable patients with acute pulmonary embolism: a prospective validation study. Circulation. 2011 Dec 13;124(24):2716-24. doi: 10.1161/CIRCULATIONAHA.111.051177. Epub 2011 Nov 14. PMID 22082681
- [Background] Sztrymf B, Souza R, Bertoletti L, Jais X, Sitbon O, Price LC, Simonneau G, Humbert M. Prognostic factors of acute heart failure in patients with pulmonary arterial hypertension. Eur Respir J. 2010 Jun;35(6):1286-93. doi: 10.1183/09031936.00070209. Epub 2009 Nov 6. PMID 19897557
- [Background] Naito A, Tanabe N, Jujo T, Shigeta A, Sugiura T, Sakao S, Ishida K, Tatsumi K. Pentraxin3 in chronic thromboembolic pulmonary hypertension: a new biomarker for screening from remitted pulmonary thromboembolism. PLoS One. 2014 Nov 20;9(11):e113086. doi: 10.1371/journal.pone.0113086. eCollection 2014. PMID 25412085
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Ghignone M, Girling L, Prewitt RM. Volume expansion versus norepinephrine in treatment of a low cardiac output complicating an acute increase in right ventricular afterload in dogs. Anesthesiology. 1984 Feb;60(2):132-5. doi: 10.1097/00000542-198402000-00009. PMID 6198941
- [Background] Zannad F, Adamopoulos C, Mebazaa A, Gheorghiade M. The challenge of acute decompensated heart failure. Heart Fail Rev. 2006 Jun;11(2):135-9. doi: 10.1007/s10741-006-9484-x. PMID 16937032
- [Background] Ng TM, Singh AK, Dasta JF, Feldman D, Mebazaa A. Contemporary issues in the pharmacologic management of acute heart failure. Crit Care Clin. 2006 Apr;22(2):199-219, v. doi: 10.1016/j.ccc.2006.02.008. PMID 16677996
- [Background] De Luca L, Fonarow GC, Adams KF Jr, Mebazaa A, Tavazzi L, Swedberg K, Gheorghiade M. Acute heart failure syndromes: clinical scenarios and pathophysiologic targets for therapy. Heart Fail Rev. 2007 Jun;12(2):97-104. doi: 10.1007/s10741-007-9011-8. PMID 17487581
- [Background] Mebazaa A, Nieminen MS, Packer M, Cohen-Solal A, Kleber FX, Pocock SJ, Thakkar R, Padley RJ, Poder P, Kivikko M; SURVIVE Investigators. Levosimendan vs dobutamine for patients with acute decompensated heart failure: the SURVIVE Randomized Trial. JAMA. 2007 May 2;297(17):1883-91. doi: 10.1001/jama.297.17.1883. PMID 17473298
- [Background] Adamopoulos C, Zannad F, Fay R, Mebazaa A, Cohen-Solal A, Guize L, Juilliere Y, Alla F. Ejection fraction and blood pressure are important and interactive predictors of 4-week mortality in severe acute heart failure. Eur J Heart Fail. 2007 Sep;9(9):935-41. doi: 10.1016/j.ejheart.2007.06.001. Epub 2007 Jul 12. PMID 17627880
- [Background] Pang PS, Cleland JG, Teerlink JR, Collins SP, Lindsell CJ, Sopko G, Peacock WF, Fonarow GC, Aldeen AZ, Kirk JD, Storrow AB, Tavares M, Mebazaa A, Roland E, Massie BM, Maisel AS, Komajda M, Filippatos G, Gheorghiade M; Acute Heart Failure Syndromes International Working Group. A proposal to standardize dyspnoea measurement in clinical trials of acute heart failure syndromes: the need for a uniform approach. Eur Heart J. 2008 Mar;29(6):816-24. doi: 10.1093/eurheartj/ehn048. Epub 2008 Mar 1. PMID 18310669
- [Background] Huvelle E, Fay R, Alla F, Cohen Solal A, Mebazaa A, Zannad F. Left bundle branch block and mortality in patients with acute heart failure syndrome: a substudy of the EFICA cohort. Eur J Heart Fail. 2010 Feb;12(2):156-63. doi: 10.1093/eurjhf/hfp180. Epub 2009 Dec 21. PMID 20028696
- [Background] Mebazaa A, Pang PS, Tavares M, Collins SP, Storrow AB, Laribi S, Andre S, Mark Courtney D, Hasa J, Spinar J, Masip J, Frank Peacock W, Sliwa K, Gayat E, Filippatos G, Cleland JG, Gheorghiade M. The impact of early standard therapy on dyspnoea in patients with acute heart failure: the URGENT-dyspnoea study. Eur Heart J. 2010 Apr;31(7):832-41. doi: 10.1093/eurheartj/ehp458. Epub 2009 Nov 11. PMID 19906690
- [Background] Bohm M, Link A, Cai D, Nieminen MS, Filippatos GS, Salem R, Cohen Solal A, Huang B, Padley RJ, Kivikko M, Mebazaa A. Beneficial association of beta-blocker therapy on recovery from severe acute heart failure treatment: data from the Survival of Patients With Acute Heart Failure in Need of Intravenous Inotropic Support trial. Crit Care Med. 2011 May;39(5):940-4. doi: 10.1097/CCM.0b013e31820a91ed. PMID 21283007
- [Background] Laribi S, Aouba A, Nikolaou M, Lassus J, Cohen-Solal A, Plaisance P, Pavillon G, Jois P, Fonarow GC, Jougla E, Mebazaa A; GREAT network. Trends in death attributed to heart failure over the past two decades in Europe. Eur J Heart Fail. 2012 Mar;14(3):234-9. doi: 10.1093/eurjhf/hfr182. Epub 2012 Jan 10. PMID 22237388
- [Background] Parissis JT, Rafouli-Stergiou P, Mebazaa A, Ikonomidis I, Bistola V, Nikolaou M, Meas T, Delgado J, Vilas-Boas F, Paraskevaidis I, Anastasiou-Nana M, Follath F. Acute heart failure in patients with diabetes mellitus: clinical characteristics and predictors of in-hospital mortality. Int J Cardiol. 2012 May 17;157(1):108-13. doi: 10.1016/j.ijcard.2011.11.098. Epub 2011 Dec 15. PMID 22178056
- [Background] Mebazaa A, Vanpoucke G, Thomas G, Verleysen K, Cohen-Solal A, Vanderheyden M, Bartunek J, Mueller C, Launay JM, Van Landuyt N, D'Hondt F, Verschuere E, Vanhaute C, Tuytten R, Vanneste L, De Cremer K, Wuyts J, Davies H, Moerman P, Logeart D, Collet C, Lortat-Jacob B, Tavares M, Laroy W, Januzzi JL, Samuel JL, Kas K. Unbiased plasma proteomics for novel diagnostic biomarkers in cardiovascular disease: identification of quiescin Q6 as a candidate biomarker of acutely decompensated heart failure. Eur Heart J. 2012 Sep;33(18):2317-24. doi: 10.1093/eurheartj/ehs162. Epub 2012 Jun 24. PMID 22733835
- [Background] Breidthardt T, Vanpoucke G, Potocki M, Mosimann T, Ziller R, Thomas G, Laroy W, Moerman P, Socrates T, Drexler B, Mebazaa A, Kas K, Mueller C. The novel marker LTBP2 predicts all-cause and pulmonary death in patients with acute dyspnoea. Clin Sci (Lond). 2012 Nov;123(9):557-66. doi: 10.1042/CS20120058. PMID 22587491
- [Background] Mebazaa A, Gayat E, Lassus J, Meas T, Mueller C, Maggioni A, Peacock F, Spinar J, Harjola VP, van Kimmenade R, Pathak A, Mueller T, Tavazzi L, Disomma S, Metra M, Pascual-Figal D, Laribi S, Logeart D, Nouira S, Sato N, Parenica J, Deye N, Boukef R, Collet C, Van den Berghe G, Cohen-Solal A, Januzzi JL Jr; GREAT Network. Association between elevated blood glucose and outcome in acute heart failure: results from an international observational cohort. J Am Coll Cardiol. 2013 Feb 26;61(8):820-9. doi: 10.1016/j.jacc.2012.11.054. Epub 2013 Jan 16. PMID 23333145
- [Background] Lassus J, Gayat E, Mueller C, Peacock WF, Spinar J, Harjola VP, van Kimmenade R, Pathak A, Mueller T, Disomma S, Metra M, Pascual-Figal D, Laribi S, Logeart D, Nouira S, Sato N, Potocki M, Parenica J, Collet C, Cohen-Solal A, Januzzi JL Jr, Mebazaa A; GREAT-Network. Incremental value of biomarkers to clinical variables for mortality prediction in acutely decompensated heart failure: the Multinational Observational Cohort on Acute Heart Failure (MOCA) study. Int J Cardiol. 2013 Oct 3;168(3):2186-94. doi: 10.1016/j.ijcard.2013.01.228. Epub 2013 Mar 26. PMID 23538053
- [Background] Seronde MF, Gayat E, Logeart D, Lassus J, Laribi S, Boukef R, Sibellas F, Launay JM, Manivet P, Sadoune M, Nouira S, Solal AC, Mebazaa A; Great network. Comparison of the diagnostic and prognostic values of B-type and atrial-type natriuretic peptides in acute heart failure. Int J Cardiol. 2013 Oct 9;168(4):3404-11. doi: 10.1016/j.ijcard.2013.04.164. Epub 2013 May 14. PMID 23684562
- [Background] Shah R, Gayat E, Januzzi JL Jr, Sato N, Cohen-Solal A, diSomma S, Fairman E, Harjola VP, Ishihara S, Lassus J, Maggioni A, Metra M, Mueller C, Mueller T, Parenica J, Pascual-Figal D, Peacock WF, Spinar J, van Kimmenade R, Mebazaa A; GREAT (Global Research on Acute Conditions Team) Network. Body mass index and mortality in acutely decompensated heart failure across the world: a global obesity paradox. J Am Coll Cardiol. 2014 Mar 4;63(8):778-85. doi: 10.1016/j.jacc.2013.09.072. Epub 2013 Dec 4. PMID 24315906
- [Background] Cohen AT, Spiro TE, Spyropoulos AC, Desanctis YH, Homering M, Buller HR, Haskell L, Hu D, Hull R, Mebazaa A, Merli G, Schellong S, Tapson VF, Burton P; MAGELLAN Study Group. D-dimer as a predictor of venous thromboembolism in acutely ill, hospitalized patients: a subanalysis of the randomized controlled MAGELLAN trial. J Thromb Haemost. 2014 Apr;12(4):479-87. doi: 10.1111/jth.12515. PMID 24460645
- [Background] Pang PS, Collins SP, Sauser K, Andrei AC, Storrow AB, Hollander JE, Tavares M, Spinar J, Macarie C, Raev D, Nowak R, Gheorghiade M, Mebazaa A. Assessment of dyspnea early in acute heart failure: patient characteristics and response differences between likert and visual analog scales. Acad Emerg Med. 2014 Jun;21(6):659-66. doi: 10.1111/acem.12390. PMID 25039550
- [Background] Mebazaa A, Spiro TE, Buller HR, Haskell L, Hu D, Hull R, Merli G, Schellong SW, Spyropoulos AC, Tapson VF, De Sanctis Y, Cohen AT. Predicting the risk of venous thromboembolism in patients hospitalized with heart failure. Circulation. 2014 Jul 29;130(5):410-8. doi: 10.1161/CIRCULATIONAHA.113.003126. Epub 2014 Jun 26. PMID 24970782
- [Background] Vodovar N, Seronde MF, Laribi S, Gayat E, Lassus J, Boukef R, Nouira S, Manivet P, Samuel JL, Logeart D, Ishihara S, Cohen Solal A, Januzzi JL Jr, Richards AM, Launay JM, Mebazaa A; GREAT Network. Post-translational modifications enhance NT-proBNP and BNP production in acute decompensated heart failure. Eur Heart J. 2014 Dec 21;35(48):3434-41. doi: 10.1093/eurheartj/ehu314. Epub 2014 Aug 24. PMID 25157115
- [Background] Cohen-Solal A, Laribi S, Ishihara S, Vergaro G, Baudet M, Logeart D, Mebazaa A, Gayat E, Vodovar N, Pascual-Figal DA, Seronde MF. Prognostic markers of acute decompensated heart failure: the emerging roles of cardiac biomarkers and prognostic scores. Arch Cardiovasc Dis. 2015 Jan;108(1):64-74. doi: 10.1016/j.acvd.2014.10.002. Epub 2014 Nov 4. PMID 25534886
- [Background] Parissis JT, Andreoli C, Kadoglou N, Ikonomidis I, Farmakis D, Dimopoulou I, Iliodromitis E, Anastasiou-Nana M, Lainscak M, Ambrosio G, Mebazaa A, Filippatos G, Follath F. Differences in clinical characteristics, management and short-term outcome between acute heart failure patients chronic obstructive pulmonary disease and those without this co-morbidity. Clin Res Cardiol. 2014 Sep;103(9):733-41. doi: 10.1007/s00392-014-0708-0. Epub 2014 Apr 10. PMID 24718849
- [Background] Legrand M, Mebazaa A, Ronco C, Januzzi JL Jr. When cardiac failure, kidney dysfunction, and kidney injury intersect in acute conditions: the case of cardiorenal syndrome. Crit Care Med. 2014 Sep;42(9):2109-17. doi: 10.1097/CCM.0000000000000404. PMID 24810531
- [Background] Kelly JP, Mentz RJ, Mebazaa A, Voors AA, Butler J, Roessig L, Fiuzat M, Zannad F, Pitt B, O'Connor CM, Lam CSP. Patient selection in heart failure with preserved ejection fraction clinical trials. J Am Coll Cardiol. 2015 Apr 28;65(16):1668-1682. doi: 10.1016/j.jacc.2015.03.043. PMID 25908073
- [Background] Mebazaa A, Yilmaz MB, Levy P, Ponikowski P, Peacock WF, Laribi S, Ristic AD, Lambrinou E, Masip J, Riley JP, McDonagh T, Mueller C, deFilippi C, Harjola VP, Thiele H, Piepoli MF, Metra M, Maggioni A, McMurray J, Dickstein K, Damman K, Seferovic PM, Ruschitzka F, Leite-Moreira AF, Bellou A, Anker SD, Filippatos G. Recommendations on pre-hospital & early hospital management of acute heart failure: a consensus paper from the Heart Failure Association of the European Society of Cardiology, the European Society of Emergency Medicine and the Society of Academic Emergency Medicine. Eur J Heart Fail. 2015 Jun;17(6):544-58. doi: 10.1002/ejhf.289. Epub 2015 May 21. PMID 25999021
- [Background] Mebazaa A, Longrois D, Metra M, Mueller C, Richards AM, Roessig L, Seronde MF, Sato N, Stockbridge NL, Gattis Stough W, Alonso A, Cody RJ, Cook Bruns N, Gheorghiade M, Holzmeister J, Laribi S, Zannad F. Agents with vasodilator properties in acute heart failure: how to design successful trials. Eur J Heart Fail. 2015 Jul;17(7):652-64. doi: 10.1002/ejhf.294. Epub 2015 Jun 4. PMID 26040488
- [Background] Jaffe AS, Apple FS, Mebazaa A, Vodovar N. Unraveling N-terminal pro-B-type natriuretic peptide: another piece to a very complex puzzle in heart failure patients. Clin Chem. 2015 Aug;61(8):1016-8. doi: 10.1373/clinchem.2015.243626. Epub 2015 Jun 15. No abstract available. PMID 26078443
- [Background] Gayat E, Caillard A, Laribi S, Mueller C, Sadoune M, Seronde MF, Maisel A, Bartunek J, Vanderheyden M, Desutter J, Dendale P, Thomas G, Tavares M, Cohen-Solal A, Samuel JL, Mebazaa A. Soluble CD146, a new endothelial biomarker of acutely decompensated heart failure. Int J Cardiol. 2015 Nov 15;199:241-7. doi: 10.1016/j.ijcard.2015.07.039. Epub 2015 Jul 12. PMID 26209827
- [Background] Vodovar N, Seronde MF, Laribi S, Gayat E, Lassus J, Januzzi JL Jr, Boukef R, Nouira S, Manivet P, Samuel JL, Logeart D, Cohen-Solal A, Richards AM, Launay JM, Mebazaa A; GREAT Network. Elevated Plasma B-Type Natriuretic Peptide Concentrations Directly Inhibit Circulating Neprilysin Activity in Heart Failure. JACC Heart Fail. 2015 Aug;3(8):629-36. doi: 10.1016/j.jchf.2015.03.011. PMID 26251090
- [Background] Teixeira A, Parenica J, Park JJ, Ishihara S, AlHabib KF, Laribi S, Maggioni A, Miro O, Sato N, Kajimoto K, Cohen-Solal A, Fairman E, Lassus J, Mueller C, Peacock WF, Januzzi JL Jr, Choi DJ, Plaisance P, Spinar J, Mebazaa A, Gayat E; GREAT (Global Research on Acute Conditions Team) Network. Clinical presentation and outcome by age categories in acute heart failure: results from an international observational cohort. Eur J Heart Fail. 2015 Nov;17(11):1114-23. doi: 10.1002/ejhf.330. Epub 2015 Sep 30. PMID 26419908
- [Background] Spinar J, Jarkovsky J, Spinarova L, Mebazaa A, Gayat E, Vitovec J, Linhart A, Widimsky P, Miklik R, Zeman K, Belohlavek J, Malek F, Felsoci M, Kettner J, Ostadal P, Cihalik C, Vaclavik J, Taborsky M, Dusek L, Littnerova S, Parenica J. AHEAD score--Long-term risk classification in acute heart failure. Int J Cardiol. 2016 Jan 1;202:21-6. doi: 10.1016/j.ijcard.2015.08.187. Epub 2015 Aug 28. PMID 26386914
- [Background] Mebazaa A, Tolppanen H, Mueller C, Lassus J, DiSomma S, Baksyte G, Cecconi M, Choi DJ, Cohen Solal A, Christ M, Masip J, Arrigo M, Nouira S, Ojji D, Peacock F, Richards M, Sato N, Sliwa K, Spinar J, Thiele H, Yilmaz MB, Januzzi J. Acute heart failure and cardiogenic shock: a multidisciplinary practical guidance. Intensive Care Med. 2016 Feb;42(2):147-63. doi: 10.1007/s00134-015-4041-5. Epub 2015 Sep 14. PMID 26370690
- [Background] Parissis J, Farmakis D, Kadoglou N, Ikonomidis I, Fountoulaki E, Hatziagelaki E, Deftereos S, Follath F, Mebazaa A, Lekakis J, Filippatos G. Body mass index in acute heart failure: association with clinical profile, therapeutic management and in-hospital outcome. Eur J Heart Fail. 2016 Mar;18(3):298-305. doi: 10.1002/ejhf.489. Epub 2016 Jan 28. PMID 26817848
- [Background] Harjola VP, Mebazaa A, Celutkiene J, Bettex D, Bueno H, Chioncel O, Crespo-Leiro MG, Falk V, Filippatos G, Gibbs S, Leite-Moreira A, Lassus J, Masip J, Mueller C, Mullens W, Naeije R, Nordegraaf AV, Parissis J, Riley JP, Ristic A, Rosano G, Rudiger A, Ruschitzka F, Seferovic P, Sztrymf B, Vieillard-Baron A, Yilmaz MB, Konstantinides S. Contemporary management of acute right ventricular failure: a statement from the Heart Failure Association and the Working Group on Pulmonary Circulation and Right Ventricular Function of the European Society of Cardiology. Eur J Heart Fail. 2016 Mar;18(3):226-41. doi: 10.1002/ejhf.478. PMID 26995592
- [Background] Van Aelst LN, Celutkiene J, Mebazaa A. Advanced heart failure: look right to prognosticate right! Eur J Heart Fail. 2016 May;18(5):573-5. doi: 10.1002/ejhf.533. No abstract available. PMID 27135771